CLINICAL TRIAL: NCT05892068
Title: Window of Opportunity Analysis of Pre-Operative Tucatinib for Surgically Resected HER2+ Brain Metastases: Understanding Mechanisms of Resistance
Brief Title: A Study of Tucatinib Given Before Surgery to People With HER2+ Cancers That Have Spread to the Brain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pfizer (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-168
Record Dates: First submitted 2023-05-18; First posted 2023-06-07 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Tucatinib; HER2+; Surgery; 22-168
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib

STUDY DESIGN:
Intervention Model Description: The study design includes patient candidates for clinically indicated craniotomy in three parallel cohorts.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients already on Tucatinib (Experimental): Cohort A: This is a non-interventional study patients who will enter while already on Tucatinib . Patients in cohort A who are already on Tucatinib at a dose reduction (i.e., for toxicity) will continue the same dose.
  Interventions: Drug: Tucatinib
- Patients with documented radiological and/or clinical CNS progression with no prior tucatinib (Experimental): Cohort B: Is to administer Tucatinib at standard dose of 300mg orally twice daily for 4 days prior to surgery (day -4 to 0).
  Interventions: Drug: Tucatinib
- HER2+ esophagogastric, lung, or colon cancer brain metastases and HER2 mutant breast cancer (Experimental): Cohort C: Is to administer Tucatinib at standard dose of 300mg orally twice daily for 4 days prior to surgery (day -4 to 0).
  Interventions: Drug: Tucatinib

INTERVENTIONS:
Drug: Tucatinib — Standard dose of 300mg orally twice daily for 4 days prior to surgery (day -4 to 0).

SUMMARY:
The purpose of this study to see how the brain absorbs, distributes, and gets rid of tucatinib in people who have HER2+ cancers (breast cancer, NSCLC, CRC, or GEC) that have spread to the brain, and to learn more about how cancer cells develop resistance to treatment. The researchers will do research tests to look for genetic differences between HER2+ breast cancer that has spread to the brain and progressed during treatment with tucatinib and cancers that are being treated with tucatinib for the first time.

DETAILED DESCRIPTION:
All patients will receive tucatinib per-protocol at standard dose of 300 mg orally twice daily on days - 4, -3, -2, -1 and day 0 (in AM). The post-surgery treatment (systemic and/or local) will be decided according to treating physician discretion and is not a study intervention. Tissue samples of brain metastases along with blood/plasma and CSF samples will be analyzed to evaluate brain tumor penetration of tucatinib as well as biologic response to tucatinib in patients with brain metastases from HER2+/mutant breast cancer who are undergoing clinically indicated brain surgery. Patients may continue tucatinib post-operatively at the discretion of the treating oncologist with monitoring as per clinical routine; this is not a study intervention for Cohort A and Cohort B. Patients on Cohort C may receive tucatinib post-operatively through the study according to physician descretion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years with no impairment in decision making capacity
* Patients with HER2 overexpressed/amplified/mutant metastatic breast/lung/esophagogastric/colorectal cancer (IHC, fluorescent in situ hybridation or sequencing-confirmed primary, brain, or other metastatic site) and one or more brain tumor(s) planned for neurosurgical resection. Other untreated brain metastases, and prior radiation (whole brain radiation therapy and/or stereotactic radiosurgery) to the index site are allowed
* Patients with concomitant leptomeningeal disease are eligible provided they have parenchymal brain metastases requiring resection.
* Life expectancy of >12 weeks.
* ECOG Performance Status (PS) of 0 to 2
* Prior treatments:

  * Cohort A: Clinical and or radiological CNS parenchymal progression on tucatinib as most recent line of treatment (tucatinib-resistant) in patients with HER2 overexpressed/amplified breast cancer
  * Clinical and or radiological CNS parenchymal progression with no prior tucatinib (tucatinib naïve) in patients with HER2 overexpressed/amplified breast cancer
  * Clinical and or radiological CNS parenchymal progression in patients with HER2+/mutant lung/esophagogastric/colorectal cancer and HER2 mutant breast cancer

ALL PATIENTS:

* Prior conventional dose lapatinib and neratinib are allowed in any cohort if > 6 months prior
* No limit on prior lines of systemic therapy
* Adequate bone marrow, liver, renal function, and coagulation parameters (obtained ≤ 7 days prior to the first day of study treatment:

  1. Absolute neutrophil count (ANC) ≥1.0 × 103μL, Platelet count ≥75 × 103 /μL, Hemoglobin ≥ 8.0 g/dL
  2. Total bilirubin ≤1.5 × upper limit of normal (ULN). Subjects with known history of Gilbert's Syndrome and normal direct bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) are eligible: AST and ALT ≤2.5 × ULN (≤5 × ULN if liver metastases are present)
  3. Calculated creatinine clearance ≥50 mL/min using the CKD-EPI (2021) (in Cohort A, in patients with elevated serum creatinine, eGFR can be calculated using cystatin C to confirm eligibility)
  4. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless on medication known to alter INR and/or aPTT
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to enrollment and must agree to use adequate contraception prior to enrollment and for the duration of study participation
* Patients must be able to swallow and retain oral medication

Exclusion Criteria:

* Contraindications or history of allergic reaction to tucatinib or any of its excipients
* Significant medical co-morbidities as per investigator evaluation
* Inability to comply with protocol and /or not willing or not available for follow-up assessments or any condition which in the investigator's opinion makes the patient unsuitable for the study participation
* Have used a strong or moderate CYP2C8 inhibitor within 5 half-lives of the inhibitor or have used a strong or moderate CYP2C8 or CYP3A4 inducer within 2 weeks prior to first dose of study treatment (Appendix E)
* Receiving concomitant CYP3A or P-gp substrates where minimal concentration changes may lead to serious or life-threatening toxicities
* Concurrent pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 28 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2028-05-09 (Estimated); Study Completion 2028-05-09 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of Tucatinib | 3 days after treatment
  by measurement of intrametastasis levels

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Seidman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm